CLINICAL TRIAL: NCT00741403
Title: An Open Label, Dose-Escalation Study to Evaluate Safety, Tolerability, Maximum Tolerated Dose (MTD), Efficacy, and Pharmacokinetics (PKs) of CPI-613 Given Twice Weekly for Three Consecutive Weeks in Cancer Patients
Brief Title: A Open Label Phase I/II Clinical Trial to Evaluate CPI-613 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cornerstone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-CPI-613-002
Record Dates: First submitted 2008-08-25; First posted 2008-08-26 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Advanced Cancer; Metastatic Cancer; Lymphoma; Solid Tumors; Advanced Malignancies
Keywords: Phase I; malignancies; refractory; relapsed
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma; Neoplasms; Recurrence | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): IV Infusion of CPI-613 on Days 1,4,8,11,15,18 of 28 day cycle in patients with advanced malignancies
  Interventions: Drug: CPI-613

INTERVENTIONS:
Drug: CPI-613 — CPI-613, the investigational drug, is a novel anti-tumor compound believed to operate via a novel mechanism of action that does not belong to any existing pharmacological class of anticancer agents currently being used in the clinics. Specifically, CPI-613 is Cornerstone Pharmaceutical Inc.'s lead drug from its Altered Energy Metabolism-Directed (AEMD) technology platform. It is selective against tumor cells (but not normal cells)according to preclinical studies

SUMMARY:
An open label, dose-escalation study to evaluate safety, tolerability, maximum tolerated dose (MTD), efficacy, and pharmacokinetics (PKs) of CPI-613 given twice weekly for three consecutive weeks in cancer patients

The objectives of this study are:

* To determine the safety and MTD of CPI-613 when administered 2x weekly for 3 consecutive weeks.
* To determine pharmacokinetics of CPI-613 following intravenous (IV) administration.
* To observe the anti-tumor effects of CPI-613, if any occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have advanced and/or metastatic, histologically or cytologically documented solid tumors and lymphomas, for whom there is no available therapy shown to provide clinical benefit.
* Karnofsky Performance Status (KPS) of >70%.
* Must be ≥18 years of age.
* Expected survival >3 months.
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device), and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation. (Note: Pregnant patients are excluded because the effects of CPI-613 on a fetus are unknown.)
* Fertile men must practice effective contraceptive methods during the study period, unless documentation of infertility exists.
* Mentally competent, ability to understand and willingness to sign the informed consent form.
* No radiotherapy, treatment with cytotoxic agents (except CPI-613), or treatment with biologic agents within the 3 weeks prior to treatment with CPI-613. At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤Grade 1 are eligible, but must be documented as such.
* Laboratory values ≤2 weeks must be:

  * Adequate hematologic (white blood cell [WBC] ≥3500 cells/mm^3 or ≥3.5 bil/L; platelet count ≥100,000 cells/mm^3 or ≥100 bil/L; absolute neutrophil count [ANC] ≥1500 cells/mm^3 or ≥1.5 bil/L; and hemoglobin (Hgb) ≥9 g/dL or ≥90 g/L).
  * Adequate hepatic function (aspartate aminotransferase [AST/SGOT] ≤3x upper normal limit [UNL], alanine aminotransferase [ALT/SGPT] ≤3x UNL (≤5x UNL if liver metastases present), bilirubin ≤1.5x UNL).
  * Adequate renal function (serum creatinine ≤2.0 mg/dL or 177 µmol/L).
  * Adequate coagulation (International Normalized Ratio or INR must be ≤1.25).

Exclusion Criteria:

* Serious medical illness, such as significant cardiac disease (symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, or New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity.
* Patients with active central nervous system (CNS) or epidural tumor.
* Any active uncontrolled bleeding, and any patients with a bleeding diathesis (e.g., active peptic ulcer disease).
* Pregnant women, or women of child-bearing potential not using reliable means of contraception (because the teratogenic potential of CPI-613 is unknown).
* Lactating females because the potential of excretion of CPI-613 into breast milk. (Note: Lactating females are excluded because the effects of CPI-613 on a nursing child are unknown.)
* Fertile men unwilling to practice contraceptive methods during the study period.
* Life expectancy less than 3 months.
* Any condition or abnormality which may, in the opinion of the investigator, compromise the safety of patients.
* Unwilling or unable to follow protocol requirements.
* Dyspnea with minimal to moderate exertion. Patients with large and recurrent pleural, or peritoneal effusions requiring frequent drainage (e.g. weekly). Patients with any amount of clinically significant pericardial effusion.
* Active heart disease including myocardial infarction within previous 6 months, symptomatic coronary artery disease, arrhythmias requiring medication, or symptomatic congestive heart failure.
* Albumin <2.5 g/dL or <25 g/L.
* Evidence of active infection, or serious infection within the past month.
* Patients with known HIV infection.
* Patients receiving any other standard or investigational treatment for their cancer, or any other investigational agent for any indication within the past 3 weeks prior to initiation of CPI-613 treatment.
* Patients who have received immunotherapy of any type within the past 4 weeks prior to initiation of CPI-613 treatment.
* Requirement for immediate palliative treatment of any kind including surgery.
* Patients that have received a chemotherapy regimen with stem cell support in the previous 6 months.
* A marked baseline prolongation of QT/QTc interval (e.g., repeated exhibition of a QTc interval >470 ms.).
* A history of additional risk factors for torsade de pointes (e.g., clinically significant heart failure, hypokalemia, family history of Long QT Syndrome).
* Troponin I above institution limit of normal or Left Ventricular Ejection Fraction (LVEF) below 35%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety, tolerability, maximum tolerated dose (MTD), and efficacy pharmacokinetics of CPI-613 given twice weekly for three consecutive weeks in cancer patients | October 2010

SECONDARY OUTCOMES:
To evaluate pharmacokinetics, toxicity profile, biological activity, and anti-tumor activity of CPI-613 given twice weekly for three consecutive weeks in cancer patients | October 2010

CONTACTS AND LOCATIONS:
Overall Officials: Karen Gelmon, M.D., Principal Investigator — British Columbia Cancer Agency; Avi Retter, M.D., Principal Investigator — Eastchester Center for Cancer Care; Divis K Khaira, M.D., Principal Investigator — Pivotal Research Centers; Senzer Neil, M.D., Principal Investigator — Mary Crowley Cancer Research Centers
Locations (4):
- United States (3):
  - Pivotal Research Centers, Peoria, Arizona
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Mary Crowley Cancer Research Centers, Dallas, Texas
- British Columbia Cancer Agency, Vancouver, British Columbia, Canada